CLINICAL TRIAL: NCT00455351
Title: Phase I Study on Suberoylanilide Hydroxyamic Acid (Vorinostat) a Histone Deacetylase Inhibitor, in Palliative Radiotherapy for Advanced Tumors.
Brief Title: Vorinostat and Palliative Radiotherapy
Acronym: PRAVO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, Senior physician, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCTnumber 2006-003631-76
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Cancer; Radiotherapy
Keywords: Palliative treatment; Max. tolerable dose
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A I (Experimental): Study drug
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Increasing dosing, phase I

SUMMARY:
Phase I study. Side-effects when combined with standard palliative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic malignancy
* Palliative radiation treatment planed
* ECOG <3
* Age>18 years

Exclusion Criteria:

* Previous pelvic radiotherapy
* Uncontrolled diarrhea
* Insulin-dependent diabetes mellitus
* BMI<18.5

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-02; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
DLT | continously

CONTACTS AND LOCATIONS:
Overall Officials: Sigbjørn Smeland, MD,PhD, Study Director — Norwegian Radium Hospital
Locations (1):
- The Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Ree AH, Dueland S, Folkvord S, Hole KH, Seierstad T, Johansen M, Abrahamsen TW, Flatmark K. Vorinostat, a histone deacetylase inhibitor, combined with pelvic palliative radiotherapy for gastrointestinal carcinoma: the Pelvic Radiation and Vorinostat (PRAVO) phase 1 study. Lancet Oncol. 2010 May;11(5):459-64. doi: 10.1016/S1470-2045(10)70058-9. Epub 2010 Apr 6. PMID 20378407
- [Derived] Bratland A, Dueland S, Hollywood D, Flatmark K, Ree AH. Gastrointestinal toxicity of vorinostat: reanalysis of phase 1 study results with emphasis on dose-volume effects of pelvic radiotherapy. Radiat Oncol. 2011 Apr 8;6:33. doi: 10.1186/1748-717X-6-33. PMID 21473790